CLINICAL TRIAL: NCT00535548
Title: Effect of Hematopoietic Stem Cells in Chronic Wounds Using a Pressure Sore Model: A Pilot Study on Feasibility, Safety and Potential Effects
Brief Title: Hematopoietic Stem Cell Therapy in Chronic Wounds Using a Pressure Sore Model
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Basel, Switzerland (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 552
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Chronic Wounds; Pressure Sores; Hematopoietic Stem Cells; Wound Healing
Keywords: Chronic wounds; Pressure sores; Hematopoietic stem cells; Wound healing
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Stem cell therapy — Injection of a hematopoietic stem cell suspension (50'000 CD 34+ cells per microliter) into the wound (1 microliter per cm2 of wound surface)

SUMMARY:
Aim of the study:

Evaluation of feasibility, safety and potential effects of stem cells on chronic wounds using a pressure sore model.

Clinical relevance:

* Accelerated healing of uncomplicated wounds
* Enhanced healing of complicated (chronic, non-healing) wounds

Study design:

* Prospective controlled phase I/II study
* Cohort of 5 patients in pilot study, then reevaluation

Patients:

- Para- and tetraplegic patients with sacral pressure sores grade III-IVA according to the classification of Daniel and Seiler

Methods:

1. First surgical intervention:

* Radical debridement of pressure sore
* Bone marrow harvest from the iliac crest
* Isolation of hematopoietic stem cells, aiming to gain > 1 mio. CD 34+ cells per patient under GMP conditions

  3. Stem cell therapy (after 2 days)
* Injection of stem cells in suspension (50'000 CD 34+ cells in 100 microliter saline per cm2 of wound surface) on one half of the total wound surface and cell-free saline on the other half as a control

  4. Second surgical intervention (after 3-4 weeks):
* Complete excision of the wound
* Closure of the defect by fasciocutaneous flap

  5. Evaluation of wound healing:
* Clinical
* 3D laser imaging
* Histology
* Growth factor assay

ELIGIBILITY:
Inclusion Criteria:

* Para- or tetraplegic
* Sacral pressure sores
* Grade III-IV according to classification of Daniel and Seiler

Exclusion Criteria:

* Diabetes mellitus
* Peripheral vascular disease
* Coronary artery disease
* Smoking
* Steroids and other immunosuppressive drugs
* Systemic autoimmune or rheumatoid diseases
* HIV
* Hepatitis B/C

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2007-01; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
feasibility, safety, efficacy | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Scheufler, MD, PhD, Study Director — University Hospital Basel, Spitalstrasse 21, 4031 Basel, Switzerland
Locations (1):
- Swiss Paraplegic Center, Nottwil, Switzerland

REFERENCES:
- [Derived] Wettstein R, Savic M, Pierer G, Scheufler O, Haug M, Halter J, Gratwohl A, Baumberger M, Schaefer DJ, Kalbermatten DF. Progenitor cell therapy for sacral pressure sore: a pilot study with a novel human chronic wound model. Stem Cell Res Ther. 2014 Jan 29;5(1):18. doi: 10.1186/scrt407. PMID 24476740